CLINICAL TRIAL: NCT03089450
Title: A Multicenter, Subject-blinded, Randomized Study to Evaluate Safety and Efficacy of CGBIO Stent Compared to Biomatrix Flex Stent in Patients Undergoing Drug-eluting Stent Procedure After Coronary Angiography
Brief Title: To Evaluate Safety and Efficacy of CGBIO Stent Compared to Biomatrix Flex Stent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CGBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CG-DE-225-008
Record Dates: First submitted 2017-03-19; First posted 2017-03-24 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Ischemic Heart Disease; Stable Coronary Artery Disease; Stable Angina; Unstable Angina; NSTEMI - Non-ST Segment Elevation MI
MeSH Terms: conditions — Myocardial Ischemia; Angina, Stable; Angina, Unstable; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGBIO stent (DES) (Experimental): The Co-Cr biodegradable polymer DES Sirolimus DRUG Ascorbic Acid(Vitamin C)
  Interventions: Device: CGBio stent
- Biomatrix flex(DES) (Active Comparator): The abluminal biodegradable polymer DES BA9™ (BIOLIMUS A9™) DRUG
  Interventions: Device: Biomatrix flex

INTERVENTIONS:
Device: CGBio stent — Percutaneous Coronary Intervention
  Arms: CGBIO stent (DES)
Device: Biomatrix flex — Percutaneous Coronary Intervention
  Arms: Biomatrix flex(DES)

SUMMARY:
to evaluate safety and efficacy of CGBIO stent(DES) compared to Biomatrix flex stent(DES)

DETAILED DESCRIPTION:
A Multicenter, subject-blinded, randomized study to evaluate safety and efficacy of CGBIO stent compared to Biomatrix Flex stent in patients undergoing drug-eluting stent procedure after coronary angiography

ELIGIBILITY:
Inclusion Criteria:

* At least one lesion with a diameter stenosis >50%
* suitable for coronary stent implantation in a vessel with a reference diameter ranging from 2.5 mm to 4.0 mm;
* Gr 1 ≤TIMI flow

Exclusion Criteria:

* ST-segment elevation MI
* Bifurcation lesion
* Chronic total occulusion
* Restenosis lesion
* Graft vessel lesion
* Patient has a history of bleeding diathesis or coagulopathy or patients in whom anti-platelet and/or anticoagulant therapy is contraindicated or in which patient will not be able to comply with dual antiplatelet therapy for at least 1 year
* Cardiogenic shock or hemodynamic compromise
* Existing impairment in liver and kidney.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2017-03-22 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
in-segment late loss | 9 month
  angiographic in-segment late loss measure by QCA program

SECONDARY OUTCOMES:
in-stent late loss | 9 month
  angiographic in-stent late loss measure by QCA program
MACE | 9 month
  death, MI and TVF
Restenosis rate | 9month
  angiographic restenosis rate

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo KIim, MD/PhD, Study Chair — Soeoul national university hospital; Young-Hyo Lim, MD/PhD, Principal Investigator — Hanyang University; Junghan Yoon, MD/PhD, Principal Investigator — Wonju Severance Christian Hospital
Locations (1):
- Soeul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No